CLINICAL TRIAL: NCT04449289
Title: Influence of Local Anesthetic Administration on the Cancer Recurrence Rate After Pancreatic Oncologic Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor (Other)
Responsible Party: Principal Investigator, Theodor Bot, PhD student, Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 43/3.02.2020
Record Dates: First submitted 2020-06-24; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous lidocaine (Active Comparator): Patients will be subjected to anesthesia with sevoflurane+fentanyl+intravenous lidocaine infusion for the first 48 hours postoperative
  Interventions: Drug: Intravenous lidocaine
- Epidural ropivacaine (Active Comparator): Patients will be subjected to anesthesia with sevoflurane+fentanyl+epidural ropivacaine infusion for the first 48 hours postoperatively
  Interventions: Drug: Epidural ropivacaine

INTERVENTIONS:
Drug: Intravenous lidocaine — Intraoperatively and postoperatively a standard intravenous infusion of lidocaine will be used for analgesia
  Arms: Intravenous lidocaine
Drug: Epidural ropivacaine — Intraoperatively and postoperatively an epidural infusion of ropivacaine will be used for analgesia
  Arms: Epidural ropivacaine

SUMMARY:
Study aims to compare the influence of intravenous lidocaine and peridural ropivacaine on postoperative long and short term outcome in patients with pancreatic cancer undergoing surgery.

As short term endpoints: postoperative complications and resumption of bowel function.

Long term endpoints include: 1 and 3 year recurrence and mortality.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of pancreatic cancer
* American Society of Anesthesiologists (ASA) risk I - III

Exclusion Criteria:

* chronic pain
* chronic medication that may interfere with pain: antiepileptics, NSAID, corticoids
* contraindications for any of the study medications
* significant psychiatric disorders (major depression, bipolar disorders, schizophrenia, etc.)
* Convulsive disorders requiring medication during the last 2 years
* liver cirrhosis/chronic kidney disease stage IV or V/chronic heart failure class III or IV/ decompensated diabetes
* Corticoid dependent asthma
* Autoimmune disorders
* Anti-arrhythmic medication (verapamil, propafenone, amiodarone) that may interfere with lidocaine's anti-arrhythmic effects
* Refusal for study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
1- and 3-years recurrence rate after surgery | 3 years
  Study participants will be contacted by study team via phone or e-mail

SECONDARY OUTCOMES:
1- and 3-years survival after surgery | 3 years
  Study participants will be contacted by study team via phone or e-mail
Lidocaine and ropivacaine concentration | Intraoperatively
Complication rate after surgery | 2 weeks
  Resumption of bowel function, anastomotic leakage or hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ionescu, MD PhD, Study Director — Regional Institute of Gastroenterology and Hepatology Prof. Dr. O. Fodor
Locations (1):
- Regional Institute of Gastroenterology and Hepatology "Prof. Dr. O. Fodor", Cluj-Napoca, Romania